CLINICAL TRIAL: NCT02813811
Title: A Prospective, Single Arm, Cohort Study of Nocturnal Temperature-controlled Laminar Airflow (TLA) Treatment (Airsonett®) in Patients With Allergic Asthma to Determine the Effect of Long-term Treatment on Exacerbation Frequency.
Brief Title: Laminar Airflow in Severe Asthma for Exacerbation Reduction - 48 Month Follow-up.
Acronym: LASER-48
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: Airsonett AB (Industry)
Responsible Party: Sponsor
Other Study IDs: PHT/2015/115
Record Dates: First submitted 2016-06-09; First posted 2016-06-27 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Asthma
Keywords: Temperature-controlled Laminar Airflow; Exacerbation frequency
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Temperature-controlled Laminar Airflow (TLA) treatment delivered by the Airsonett treatment device is a new treatment for patients with allergic asthma.

The LASER Trial (temperature-controlled Laminar Airflow in Severe asthma for Exacerbation Reduction - LASER) is a trial, currently evaluating whether the Airsonett device is able to reduce the frequency of asthma attacks in patients with allergic asthma. (www.lasertrial.co.uk)

Participants who successfully complete at least 6 months of follow-up in the LASER trial are eligible for the post trial provision of 4 years of an active TLA treatment device.

To date there is no long term performance data available to show whether there is any sustained benefit from the long term use of the Airsonett device, whether any improvement in asthma control or quality of life is maintained and whether patients will continue to use the treatment device beyond 12 months (the length of the longest previous trials of TLA treatment.)

The investigators plan to assess the performance of the Airsonett device by recording the frequency of asthma attacks in patients over a 4-year period (48 months.) The investigators also wish to evaluate the effect of long term TLA treatment on asthma control, quality of life, healthcare resource use and patient acceptability of longer term use of the Airsonett device.

Participants will be sent and asked to complete a series of questionnaires on a 6 monthly basis over the 48 month study period. Questionnaires will be returned by post to a single study centre based in Portsmouth, UK. Participants will also be contacted by telephone on a 6 monthly basis by a member of the trial team to collect information about their medication, healthcare resource use and whether they have had any asthma attacks since their last contact.

Participants will not be expected to visit the study centre during the trial.

DETAILED DESCRIPTION:
Asthma affects over 5.4 million people in the UK with nearly 500,00 experiencing severe symptoms and frequent exacerbations that are inadequately controlled with available treatments. The burden of severe asthma on the NHS is enormous accounting for 80% of total asthma cost. In 2009 there were 1131 deaths due to asthma, with those whose asthma remains poorly-controlled facing the greatest risk. Patients with severe asthma bear the greatest burden of asthma morbidity and experience more frequent and severe exacerbations which reduce their quality of life, impair their ability to work and place an enormous burden of anxiety on them and their families. There is also an increased risk of significant depression. 1 in 5 asthmatics in the UK report serious concerns that their next asthma attack will kill them. As highlighted in the 2010 Asthma UK report, 'Fighting for Breath,' these patients also face discrimination from employers, healthcare professional s and society as a whole as a result of their asthma.

Current treatments including oral corticosteroids, 'steroid-sparing' immunosuppressants and monoclonal antibody therapies are often of limited efficacy and have potentially serious side effects (steroids, immunosuppressive agents) or are prohibitively expensive (monoclonal antibodies). The adverse effects of long-term oral steroids include adrenal suppression, decreased bone mineral density, diabetes and increased cardiovascular mortality. The anti-IgE treatment Omalizumab® has been shown to reduce exacerbations by up to 50% and improve quality of life in severe allergic asthma but costs up to £26,640 per year, which is substantially more than the current annual rental cost of a TLA device (£2,088).

Patients with poorly controlled, severe, allergic asthma are left with a significant unmet clinical need and a specific requirement for cost-effective therapies which reduce systemic steroid exposure by reducing the frequency of severe exacerbations.

The Department of Health Outcomes Strategy for COPD and Asthma (2011) recognised the huge burden that poorly-controlled asthma places on people's lives and the NHS, and spelt out the political commitment to improve asthma control and reduce asthma related emergency healthcare needs and deaths. The 2013 British Thoracic Society (BTS) and Scottish Intercollegiate Guidelines Network (SIGN) national asthma guidelines and 2010 WHO consultation on severe asthma have highlighted an urgent need for research in severe asthma, acknowledging the limitations of available treatments in severe asthma and the dearth of clinical trials upon which to base management recommendations. Asthma UK emphasised in its research strategy for 2012 document that new therapies able to reduce symptoms and prevent exacerbations will improve clinical outcomes and patient well-being and reduce the cost of treating severe asthma within the NHS.

More than 70% of severe asthmatic patients are sensitised to common aeroallergens and/or moulds and the level of allergen exposure determines symptoms; those exposed to high allergen levels are at increased risk of exacerbations and hospital admissions. Domestic exposure to allergens is also known to act synergistically with viruses in sensitised patients to increase the risk and severity of exacerbations. Allergen avoidance has been widely recognised as a logical way of treating these patients . In controlled conditions, long-term allergen avoidance in sensitised asthmatics reduces airway inflammation with consequent symptomatic improvement, further supported by high-altitude, clean-air studies. Unfortunately, effective methods of allergen reduction have proved elusive, with current measures unable to reduce allergen load sufficiently to yield a consistent clinical improvement, thus leaving a significant gap in the potential strategies for reducing asthma severity through allergen reduction.

At night airborne particles are carried by a persistent convection current established by the warm body, transporting allergens from the bedding area to the breathing zone . Proof-of-concept studies have shown the TLA device reduces the total number of airborne particles >0.5μm in the breathing zone by 3000-fold (p<0.001), cat allergen exposure by 7-fold (p=0.043) and significantly reduces the increase in particles generated when turning in bed for all particle sizes . When compared to a best in class traditional air cleaners TLA is able to reduce exposure to potential allergens by a further 99%30. We postulate that this highly significant reduction in nocturnal exposure, targeted to the breathing zone, explains why TLA may succeed in an area where so many other measures, including air filters, have failed.

The TLA device when compared to placebo, has proven efficacy on asthma-related quality of life and bronchial inflammation (measured by exhaled nitric oxide) in a pan European multicentre Phase III study , (n=282, age range 7-70 years). The greatest benefit was seen in the more severe asthma patients requiring higher intensity treatment (GINA Steps 4-5) and in patients with poorly controlled asthma (Asthma Control Test <18). GINA Steps 4-5 are consistent with BTS/SIGN Guideline treatment Steps 4-5 (inhaled corticosteroid dose ≥1000µg/day beclomethasone (BDP) equivalent plus an additional controller medication such as a long acting ß2-agonist, leukotriene receptor antagonist or a sustained release theophylline). Whilst not powered to ascertain an effect on exacerbations, a post-hoc analysis showed a decreased exacerbation rate in more severe patients treated with TLA when compared with placebo with a trend towards significance (mean 0.23 TLA; 0.57 placebo p=0.07). A cost-effectiveness analysis based on the results from this trial also found no significant differences in ED visits, hospitalisation days, medication usage, and therefore overall costs between the two study groups . This lack of significant findings probably reflected the fact that the trial was not powered to detect differences in exacerbations, a predictor of increased asthma healthcare resource use and costs . Despite the lack of a significant reduction in healthcare resource use and associated costs, subsequent economic modelling showed that TLA would be cost-effective in Sweden at the current monthly rental price (SEK 2,000, ≈ £167), mainly due to increases in quality of life.

In order to address this important research question in severe allergic asthma, The LASER Trial, a multi-centre, randomised, double blind, placebo-controlled, parallel group trial is currently assessing whether nocturnal use of the TLA treatment device Airsonett® is able to reduce the frequency of severe asthma exacerbations in patients with poorly controlled, severe, allergic asthma. The LASER Trial received funding from the National Institute for Health Research Health Technology Assessment Programme.

In the LASER Trial, participants receive 12 months of treatment. Half of the participants receive an active TLA device and half receive a device which has been deactivated (a 'placebo' device.) Neither the patients nor researchers will know which device an individual participant has received. All participants who complete at least 6 months of follow-up within the LASER trial will be eligible for treatment with an active TLA device for 4 years regardless of whether they received an active or placebo device during the trial.

LASER-48 is the follow on study from The LASER Trial where the investigators will ask participants to continue to report their asthma attacks and symptoms during a 4 year (48-month) follow-up period by means of questionnaires to monitor whether the treatment device has an impact on their asthma symptoms and quality of life.

To reduce the burden on study participants, they will not be required to visit a hospital clinic for follow-up appointments but they will be contacted on a 6 monthly basis to gather information about their asthma symptoms, their asthma medications and whether they have been required to visit their GP or hospital for their asthma.

Participants will be free to withdraw from the study at any time without giving a reason for doing so.

At the end of the study after the last participant has completed their 48 months of follow-up, the data will be analysed to help determine whether longer term treatment with the TLA (Airsonett) device is able to reduce the frequency of asthma attacks, improve asthma symptoms, improve asthma related quality of life and remain a cost-effective and acceptable treatment for patients with severe allergic asthma.

ELIGIBILITY:
Inclusion Criteria:

The participant must meet ALL of the following criteria to be considered eligible for the study:

* Male or Female, aged 16 years or above.
* Using the TLA treatment device, Airsonett®, for the treatment of asthma.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

• Unable to comprehend the study and provide informed consent, e.g. insufficient command of English in the absence of someone to adequately interpret.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 3 populations of adults (aged ≥16yrs) with allergic asthma will be invited to participate:
  1. Patients receiving TLA treatment as part of the 4-year post trial provision period following participation in The LASER Trial where they were in the active treatment study group.
  2. Patients receiving TLA treatment as part of the 4-year post trial provision period following participation in The LASER Trial where they were in the placebo treatment study group.
  3. Patients starting TLA treatment for asthma who did not participate in The LASER Trial.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Frequency of severe asthma exacerbations over the 48-month follow up period. | 48 months
  Severe asthma exacerbations are defined in accordance with ATS/ERS guidelines as a worsening of asthma requiring systemic corticosteroids, ≥30mg prednisolone or equivalent daily (or ≥50% increase in dose if maintenance 30mg prednisolone or above) for 3 or more days. Courses of corticosteroids separated by ≥7 days will be treated as separate severe exacerbations.
  Participants will keep a record of their asthma exacerbations. They will be asked to record systemic corticosteroid use, dose of systemic corticosteroids and length of treatment course. This information will be collected from participants at 6, 12, 18, 24, 30, 36, 42 and 48 months.

SECONDARY OUTCOMES:
Current asthma control | 6, 12, 18, 24, 30, 36, 42 and 48 months
  Current asthma control will be recorded at 6, 12, 18, 24, 30, 36, 42 and 48 months.
  This will be measured using the Asthma Control Questionnaire.
Exacerbation Frequency | 48 months
  Risk of adverse asthma outcomes will be recorded over the 48 month study period at 6, 12, 18, 24, 30, 36, 42 and 48 months
Oral Corticosteroid Use | 6, 12, 18, 24, 30, 36, 42 and 48 months
  Risk of adverse asthma outcomes will be recorded over the 48 month study period at 6, 12, 18, 24, 30, 36, 42 and 48 months
Frequency of Hospital Admissions for Asthma | 6, 12, 18, 24, 30, 36, 42 and 48 months
  Risk of adverse asthma outcomes will be recorded over the 48 month study period at 6, 12, 18, 24, 30, 36, 42 and 48 months
Health Related Quality of Life - Mini Asthma Quality of Life Questionnaire | 6, 12, 18, 24, 30, 36, 42 and 48 months
  This will be measured using the mini Asthma Quality of Life Questionnaire (miniAQLQ) at 6, 12, 18, 24, 30, 36, 42 and 48 months.
Health Related Quality of Life - EQ-5D-5L health questionnaire | 6, 12, 18, 24, 30, 36, 42 and 48 months
  This will also be measured using the the EQ-5D-5L health questionnaire at 6, 12, 18, 24, 30, 36, 42 and 48 months.
Sino-nasal Symptoms | 6, 12, 18, 24, 30, 36, 42 and 48 months
  This will be measured using the SNOT-22 (Sino-Nasal Outcome Test questionnaire at 6, 12, 18, 24, 30, 36, 42 and 48 months.
Health Economics | 48 months
  Healthcare resource use and cost will be measured and participants will complete the Work Productivity and Activity Impairment (WPAI(A)) Questionnaire.
TLA Treatment Acceptability | 12, 24, 36 and 48 months
  Time to withdrawal of treatment and participants perception of the TLA device will be recorded at 12, 24, 36 and 48 months.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Anoop J Chauhan, MB ChB, MRCP, Principal Investigator — Consultant Respiratory Physician and Director of Research & Innovation
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bousquet J, Mantzouranis E, Cruz AA, Ait-Khaled N, Baena-Cagnani CE, Bleecker ER, Brightling CE, Burney P, Bush A, Busse WW, Casale TB, Chan-Yeung M, Chen R, Chowdhury B, Chung KF, Dahl R, Drazen JM, Fabbri LM, Holgate ST, Kauffmann F, Haahtela T, Khaltaev N, Kiley JP, Masjedi MR, Mohammad Y, O'Byrne P, Partridge MR, Rabe KF, Togias A, van Weel C, Wenzel S, Zhong N, Zuberbier T. Uniform definition of asthma severity, control, and exacerbations: document presented for the World Health Organization Consultation on Severe Asthma. J Allergy Clin Immunol. 2010 Nov;126(5):926-38. doi: 10.1016/j.jaci.2010.07.019. PMID 20926125
- [Background] Holgate ST, Polosa R. The mechanisms, diagnosis, and management of severe asthma in adults. Lancet. 2006 Aug 26;368(9537):780-93. doi: 10.1016/S0140-6736(06)69288-X. PMID 16935689
- [Background] Hoskins G, McCowan C, Neville RG, Thomas GE, Smith B, Silverman S. Risk factors and costs associated with an asthma attack. Thorax. 2000 Jan;55(1):19-24. doi: 10.1136/thorax.55.1.19. PMID 10607797
- [Background] Tough SC, Hessel PA, Ruff M, Green FH, Mitchell I, Butt JC. Features that distinguish those who die from asthma from community controls with asthma. J Asthma. 1998;35(8):657-65. doi: 10.3109/02770909809048968. PMID 9860086
- [Background] Turner MO, Noertjojo K, Vedal S, Bai T, Crump S, Fitzgerald JM. Risk factors for near-fatal asthma. A case-control study in hospitalized patients with asthma. Am J Respir Crit Care Med. 1998 Jun;157(6 Pt 1):1804-9. doi: 10.1164/ajrccm.157.6.9708092. PMID 9620909
- [Background] Campbell MJ, Holgate ST, Johnston SL. Trends in asthma mortality. Data on seasonality of deaths due to asthma were omitted from paper but editorial's author did not know. BMJ. 1997 Oct 18;315(7114):1012. No abstract available. PMID 9365305
- [Background] Rodrigo GJ, Rodrigo C, Hall JB. Acute asthma in adults: a review. Chest. 2004 Mar;125(3):1081-102. doi: 10.1378/chest.125.3.1081. PMID 15006973
- [Background] Nejtek VA, Brown ES, Khan DA, Moore JJ, Van Wagner J, Perantie DC. Prevalence of mood disorders and relationship to asthma severity in patients at an inner-city asthma clinic. Ann Allergy Asthma Immunol. 2001 Aug;87(2):129-33. doi: 10.1016/s1081-1206(10)62206-5. PMID 11527244
- [Background] Manson SC, Brown RE, Cerulli A, Vidaurre CF. The cumulative burden of oral corticosteroid side effects and the economic implications of steroid use. Respir Med. 2009 Jul;103(7):975-94. doi: 10.1016/j.rmed.2009.01.003. Epub 2009 Apr 15. PMID 19372037
- [Background] Humbert M, Beasley R, Ayres J, Slavin R, Hebert J, Bousquet J, Beeh KM, Ramos S, Canonica GW, Hedgecock S, Fox H, Blogg M, Surrey K. Benefits of omalizumab as add-on therapy in patients with severe persistent asthma who are inadequately controlled despite best available therapy (GINA 2002 step 4 treatment): INNOVATE. Allergy. 2005 Mar;60(3):309-16. doi: 10.1111/j.1398-9995.2004.00772.x. PMID 15679715
- [Background] Heaney LG, Brightling CE, Menzies-Gow A, Stevenson M, Niven RM; British Thoracic Society Difficult Asthma Network. Refractory asthma in the UK: cross-sectional findings from a UK multicentre registry. Thorax. 2010 Sep;65(9):787-94. doi: 10.1136/thx.2010.137414. PMID 20805172
- [Background] Custovic A, Taggart SC, Francis HC, Chapman MD, Woodcock A. Exposure to house dust mite allergens and the clinical activity of asthma. J Allergy Clin Immunol. 1996 Jul;98(1):64-72. doi: 10.1016/s0091-6749(96)70227-0. PMID 8765819
- [Background] Tunnicliffe WS, Fletcher TJ, Hammond K, Roberts K, Custovic A, Simpson A, Woodcock A, Ayres JG. Sensitivity and exposure to indoor allergens in adults with differing asthma severity. Eur Respir J. 1999 Mar;13(3):654-9. doi: 10.1183/09031936.99.13365499. PMID 10232442
- [Background] Langley SJ, Goldthorpe S, Craven M, Morris J, Woodcock A, Custovic A. Exposure and sensitization to indoor allergens: association with lung function, bronchial reactivity, and exhaled nitric oxide measures in asthma. J Allergy Clin Immunol. 2003 Aug;112(2):362-8. doi: 10.1067/mai.2003.1654. PMID 12897743
- [Background] Rosenstreich DL, Eggleston P, Kattan M, Baker D, Slavin RG, Gergen P, Mitchell H, McNiff-Mortimer K, Lynn H, Ownby D, Malveaux F. The role of cockroach allergy and exposure to cockroach allergen in causing morbidity among inner-city children with asthma. N Engl J Med. 1997 May 8;336(19):1356-63. doi: 10.1056/NEJM199705083361904. PMID 9134876
- [Background] Green RM, Custovic A, Sanderson G, Hunter J, Johnston SL, Woodcock A. Synergism between allergens and viruses and risk of hospital admission with asthma: case-control study. BMJ. 2002 Mar 30;324(7340):763. doi: 10.1136/bmj.324.7340.763. PMID 11923159
- [Background] Custovic A, Simpson A, Chapman MD, Woodcock A. Allergen avoidance in the treatment of asthma and atopic disorders. Thorax. 1998 Jan;53(1):63-72. doi: 10.1136/thx.53.1.63. No abstract available. PMID 9577525
- [Background] van Velzen E, van den Bos JW, Benckhuijsen JA, van Essel T, de Bruijn R, Aalbers R. Effect of allergen avoidance at high altitude on direct and indirect bronchial hyperresponsiveness and markers of inflammation in children with allergic asthma. Thorax. 1996 Jun;51(6):582-4. doi: 10.1136/thx.51.6.582. PMID 8693437
- [Background] Peroni DG, Boner AL, Vallone G, Antolini I, Warner JO. Effective allergen avoidance at high altitude reduces allergen-induced bronchial hyperresponsiveness. Am J Respir Crit Care Med. 1994 Jun;149(6):1442-6. doi: 10.1164/ajrccm.149.6.8004296.
- [Background] Grootendorst DC, Dahlen SE, Van Den Bos JW, Duiverman EJ, Veselic-Charvat M, Vrijlandt EJ, O'Sullivan S, Kumlin M, Sterk PJ, Roldaan AC. Benefits of high altitude allergen avoidance in atopic adolescents with moderate to severe asthma, over and above treatment with high dose inhaled steroids. Clin Exp Allergy. 2001 Mar;31(3):400-8. doi: 10.1046/j.1365-2222.2001.01022.x. PMID 11260151
- [Background] Gotzsche PC, Johansen HK. House dust mite control measures for asthma: systematic review. Allergy. 2008 Jun;63(6):646-59. doi: 10.1111/j.1398-9995.2008.01690.x. PMID 18445182
- [Background] Sublett JL. Effectiveness of air filters and air cleaners in allergic respiratory diseases: a review of the recent literature. Curr Allergy Asthma Rep. 2011 Oct;11(5):395-402. doi: 10.1007/s11882-011-0208-5. PMID 21773748
- [Background] Boyle RJ, Pedroletti C, Wickman M, Bjermer L, Valovirta E, Dahl R, Von Berg A, Zetterstrom O, Warner JO; 4A Study Group. Nocturnal temperature controlled laminar airflow for treating atopic asthma: a randomised controlled trial. Thorax. 2012 Mar;67(3):215-21. doi: 10.1136/thoraxjnl-2011-200665. Epub 2011 Nov 30. PMID 22131290
- [Background] Schauer U, Bergmann KC, Gerstlauer M, Lehmann S, Gappa M, Brenneken A, Schulz C, Ahrens P, Schreiber J, Wittmann M, Hamelmann E; all members of the German Asthma Net (GAN). Improved asthma control in patients with severe, persistent allergic asthma after 12 months of nightly temperature-controlled laminar airflow: an observational study with retrospective comparisons. Eur Clin Respir J. 2015 Jul 29;2. doi: 10.3402/ecrj.v2.28531. eCollection 2015. PMID 26557252
- [Background] Brodtkorb TH, Zetterstrom O, Tinghog G. Cost-effectiveness of clean air administered to the breathing zone in allergic asthma. Clin Respir J. 2010 Apr;4(2):104-10. doi: 10.1111/j.1752-699X.2009.00156.x. PMID 20565484
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Juniper EF, Svensson K, Mork AC, Stahl E. Measurement properties and interpretation of three shortened versions of the asthma control questionnaire. Respir Med. 2005 May;99(5):553-8. doi: 10.1016/j.rmed.2004.10.008. Epub 2004 Nov 26. PMID 15823451
- [Background] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Background] Pickard AS, Wilke C, Jung E, Patel S, Stavem K, Lee TA. Use of a preference-based measure of health (EQ-5D) in COPD and asthma. Respir Med. 2008 Apr;102(4):519-36. doi: 10.1016/j.rmed.2007.11.016. Epub 2008 Jan 3. PMID 18180151
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- See also: Outcomes Statergy for COPD and Asthma in England (2011) - Department of Health — http://www.gov.uk/government/uploads/system/uploads/attachment_data/file/216531/dh_134001.pdf